CLINICAL TRIAL: NCT02085993
Title: A Cross-sectional Study of Patients With Immune Thrombocytopenic Purpura and Caregivers to Estimate the Proportion Who Administer Romiplostim Correctly After Receipt of Home Administration Training Materials
Brief Title: Study of Patients With ITP Estimating the Proportion Administering Romiplostim Correctly After Receiving Home Administration Training
Status: Completed | Type: Observational
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: 20120269
Record Dates: First submitted 2014-03-11; First posted 2014-03-13 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2015-12

CONDITIONS: Immune Thrombocytopenic Purpura
Keywords: romiplostim,; Nplate,; immune thrombocytopenic purpura
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- single arm: single arm study

SUMMARY:
Cross-sectional study, observation made by healthcare professionals of subjects or caregivers, administering romiplostim at their first standard-of-care visit 4 weeks after training with the home administration training pack. Further observations can also be recorded in the study if made within 16 weeks of enrolment. Data will be collected from the subjects' dose diary at their first standard of care visit to ensure there were no problems with administration while not at the clinic.

DETAILED DESCRIPTION:
This cross-sectional study involves direct observation by a healthcare professional of a series of subjects and caregivers in the act of administering romiplostim at their first standard-of-care visit occurring 4 weeks after training with the HAT pack. Further observations, if they occur, will also be recorded in the study if made within 16 weeks of enrolment. (Additional observations are voluntary and are not required for study participation; they occur only if the healthcare professional requests them.) Additionally, data will be collected from the subjects' dose diary at the first standard of care visit to ensure there were no problems with administration while not at the clinic.

ELIGIBILITY:
Inclusion Criteria:

* (1) adult ITP patient, treated per EU Summary of product characteristics (SmPC), or caregiver new (or at least a 3 month gap) to administering romiplostim,
* (2) has received HAT pack training,
* (3) available at standard-of-care medical visit 4 weeks (range 2 to 8 weeks) after HAT pack training,
* (4) patient provides informed consent.

Exclusion Criteria:

-No exclusion criteria for this observational study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ITP patients being treated with romiplostim will be approached for possible study participation. At each participating site, patients that meet the following criteria will be enrolled as a study subject. Adult ITP patients, treated per EU Summary of product characteristics (SmPC), or caregiver new (or at least a 3 month gap) to administering romiplostim, that has received HAT pack training and is available at a standard-of-care medical visit 4 weeks (range 2 to 8 weeks) after HAT pack training, the patient provides informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2014-07; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Successful self administration of romiplostim | First Standard of Care visit post Home Administration Training (range 2-8 weeks)
  to estimate the proportion of subjects and caregivers who administer romiplostim correctly after being trained with the HAT pack.

SECONDARY OUTCOMES:
successful reconstitution of romiplostim | First standard of care visit post Home Administration Training (range 2-8 weeks). Follow up visits (up to 16 weeks post enrolment)
  A yes/no indicator of whether the subject or caregiver reconstitutes romiplostim correctly.
Accuracy in administering the prescribed dose of romiplostim | First standard of care visit post Home Administration Training (range 2-8 weeks). Follow up visits (up to 16 weeks post enrolment)
  The difference between the prescribed and administered dose of romiplostim, expressed as a %.
Injects romiplostim | First standard of care visit post Home Administration Training (range 2-8 weeks). Follow up visits (up to 16 weeks post enrolment)
  A yes/no indicator of whether the subject or caregiver injects romiplostim successfully.
Administers romiplostim | Follow up visits (up to 16 weeks post enrolment)
  A yes/no indicator of whether the subject or caregiver administers romiplostim correctly.

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (21):
- Austria (2):
  - Research Site, Innsbruck
  - Research Site, Leoben
- Belgium (2):
  - Research Site, Bruges
  - Research Site, Ghent
- France (5):
  - Research Site, Créteil
  - Research Site, Limoges
  - Research Site, Montpellier
  - Research Site, Paris
  - Research Site, Pessac
- Germany (2):
  - Research Site, Berlin
  - Research Site, Kronach
- Greece (3):
  - Research Site, Athens
  - Research Site, Kalamata
  - Research Site, Thessaloniki
- Netherlands (2):
  - Research Site, The Hague
  - Research Site, Veldhoven
- Spain (3):
  - Research Site, Ávila, Castille and León
  - Research Site, Madrid, Madrid
  - Research Site, Majadahonda, Madrid
- United Kingdom (2):
  - Research Site, Leicester
  - Research Site, London

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com